CLINICAL TRIAL: NCT02118363
Title: Proof of Concept Study of the INTERACTION Technology, Monitoring of Stroke Patients in Hospital and Home Environment
Brief Title: INTERACTION, Monitoring of Stroke Patients in Hospital and Home Environment
Acronym: INTERACTION
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: University of Twente (Other); University of Pisa (Other); Roessingh (Unknown); XSens technologies B.V. (Unknown); Smartex S.r.l. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 13101; seventh framework programme (Other Grant/Funding Number: 287351)
Record Dates: First submitted 2014-04-08; First posted 2014-04-21 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Stroke
Keywords: upper limb; lower limb; monitoring; assessment; sensor
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Clinical assessment and monitoring of balance and arm function in stroke patients with sensor based measurement, in clinical and home environment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 or above
* Previous Stroke in the personal history
* Able to walk 10 meters. A walking aid (unilateral or bilateral) is permitted
* Able to walk without special shoes
* Able to raise the arm against gravity
* Able to read and understand questionnaires and able to execute commands
* Able and willing to participate in the study
* Singed Informed Consent

Exclusion Criteria:

* Contraindications on ethical grounds (vulnerable persons)
* known or suspected non-compliance, drug or alcohol abuse,
* Severe aphasia
* Severe dementia
* Severe depression
* Relevant medical disease or increased risk of rehospitalization
* Severe sensory deficits
* Severe neglect

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subakut or chronic stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2014-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
proof of concept | 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Cereneo, Vitznau, Switzerland

REFERENCES:
- [Derived] Held JPO, Klaassen B, Eenhoorn A, van Beijnum BF, Buurke JH, Veltink PH, Luft AR. Inertial Sensor Measurements of Upper-Limb Kinematics in Stroke Patients in Clinic and Home Environment. Front Bioeng Biotechnol. 2018 Apr 12;6:27. doi: 10.3389/fbioe.2018.00027. eCollection 2018. PMID 29707537
- See also: Related Info — http://cms.interaction4stroke.eu